CLINICAL TRIAL: NCT00711412
Title: A Phase II Study of Capecitabine and Oxaliplatin With Radiation for Esophageal and Gastroesophageal Junction Adenocarcinoma
Brief Title: Capecitabine, Oxaliplatin, and Radiation Therapy in Treating Patients With Esophageal or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 05I2; STU00006779 (Other: Northwestern University IRB)
Record Dates: First submitted 2008-07-05; First posted 2008-07-08 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Induction, Combination and surgery (Experimental): Weeks 1-6:
  Capecitabine 1000mg/m2 twice daily Oxaliplatin 70mg/m2 on days 1 and 8
  Weeks 7-12:
  Capecitabine 825 mg/m2 twice daily Oxaliplatin 50mg/m2 weekly Radiation 1.8 Gy Monday-Friday
  Evaluation for response and resection surgery
  Interventions: Drug: Induction Therapy - Capecitabine; Drug: Induction Therapy - Oxaliplatin; Drug: Combination Therapy - Capecitabine; Drug: Combination Therapy - Oxaliplatin; Radiation: Combination Therapy - Radiation; Procedure: Evaluation for response and surgery

INTERVENTIONS:
Drug: Induction Therapy - Capecitabine — Two 21-day cycles will be given as induction. Capecitabine will be given at 1000 mg/m2 twice daily approximately 12 hours apart for 14 days, followed by seven days off.
Drug: Induction Therapy - Oxaliplatin — Two 21-day cycles will be given as induction. Oxaliplatin will be given at 70 mg/m2 intravenously in 5% dextrose over two hours on days 1 and 8 of each cycle.
Drug: Combination Therapy - Capecitabine — Two 21-day cycles will be given for combination therapy. Capecitabine will be given at 825 mg/m2 twice daily approximately 12 hours apart for five days (Monday through Friday) followed by two days off for 51/2 weeks.
Drug: Combination Therapy - Oxaliplatin — Two 21-day cycles will be given. Oxaliplatin will be given at 50 mg/m2 intravenously in 5% dextrose over two hours on days 1, 8 and 15 of each cycle.
Radiation: Combination Therapy - Radiation — 1.8 Gy daily Monday through Friday to a total of 50.4 Gy for 6 weeks during combination therapy.
Procedure: Evaluation for response and surgery — Four to eight weeks following the completion of therapy subjects will undergo evaluation for response and surgical resection.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well giving capecitabine and oxaliplatin together with radiation therapy works in treating patients with esophageal or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the pathologic complete response in patients with adenocarcinoma of the esophagus or gastroesophageal junction treated with neoadjuvant therapy comprising capecitabine, oxaliplatin, and radiotherapy.

Secondary

* Determine the clinical response rate in patients treated with this regimen.
* Determine the recurrence rate, time to progression, and patterns of failure in patients treated with this regimen.
* Characterize the toxicity profile of this regimen in these patients.

OUTLINE:

* Induction therapy: Patients receive oral capecitabine twice daily on days 1-14 and oxaliplatin IV over 2 hours on days 1 and 8. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
* Combination chemoradiotherapy: Patients then receive oxaliplatin IV over 2 hours once weekly for 6 weeks. Patients also receive concurrent oral capecitabine twice daily and undergo radiotherapy once daily 5 days a week for 5½ weeks in the absence of disease progression or unacceptable toxicity.
* Surgery: Patients undergo surgical resection at 4-8 weeks after completion of chemoradiotherapy.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the esophagus or gastroesophageal junction

  * Stage I-IVA disease
* No distant metastatic disease (other than regional lymph nodes)
* No evidence of CNS metastases

  * CNS metastases stable for > 3 months allowed

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Consuming ≥ 1,500 calories daily
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No pre-existing neuropathy
* No prior unanticipated severe reaction to fluoropyrimidine therapy
* No known hypersensitivity to fluorouracil
* No known DPD deficiency
* No known hypersensitivity to any of the components of oxaliplatin
* No significant active infection or other severe complicated medical illness
* No clinically significant cardiac disease (e.g., congestive heart failure, symptomatic coronary artery disease, or cardiac arrhythmias not well controlled with medication)
* No myocardial infarction within the past 12 months
* No history of uncontrolled seizures, CNS disorders, or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake
* No malabsorption syndrome
* No other active malignancy within the past 3 years except cervical carcinoma in situ or nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior participation in any investigational drug study
* No prior pelvic or thoracic radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-05-31 (Actual); Primary Completion 2009-05-29 (Actual); Study Completion 2013-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Mulcahy, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on May 31, 2006 with an accrual goal of up to 43 patients. The study was designed to enroll 13 patients initially and do an interim efficacy assessment. Accrual was suspended on July 17, 2008 for this analysis and reopened on August 12, 2008. The study was closed permanently on february 24, 2009.
Groups:
- Induction and Combination Treatment: Induction Therapy: Two 21-day cycles will be given as induction. Weeks 1-6:
  Capecitabine will be given at 1000 mg/m2 twice daily approximately 12 hours apart for 14 days, followed by seven days off.
  Oxaliplatin will be given at 70 mg/m2 intravenously in 5% dextrose over 2 hours on days 1 and 8 of each cycle.
  Combination Therapy: Two 21-day cycles will be given for combination therapy Weeks 7-12:
  Capecitabine will be given at 825 mg/m2 twice daily approximately 12 hours apart for five days (Monday through Friday) followed by two days off for 51/2 weeks.
  Oxaliplatin will be given at 50 mg/m2 intravenously in 5% dextrose over two hours on days 1, 8 and 15 of each cycle.
  Radiation: 1.8 Gy daily Monday through Friday to a total of 50.4 Gy for 6 weeks during combination therapy.
  4-6 weeks later subjects will undergo evaluation for response and surgical resection.
Period: Induction Treatment
Arm/Group | Induction and Combination Treatment
Started | 44
Registered to Study | 44
Started Induction Treatment | 43
Completed | 40
Not Completed | 4
Not completed — Death | 2
Not completed — Adverse Event | 1
Not completed — Other | 1
Period: Evaluated for Combination Treatment
Arm/Group | Induction and Combination Treatment
Started | 40
Completed | 34
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Progressive disease | 2
Period: Combination Treatment
Arm/Group | Induction and Combination Treatment
Started | 34
Completed | 33
Not Completed | 1
Not completed — Progressive Disease | 1
Period: Evaluation for Response and Surgery
Arm/Group | Induction and Combination Treatment
Started | 34 (1 patient only completed 2 cycles of therapy was evaluated and eligible for surgical resection.)
Completed | 28
Not Completed | 6
Not completed — Progressive Disease | 2
Not completed — Too high risk for surgery | 2
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Period: Survival Follow up Until Death
Arm/Group | Induction and Combination Treatment
Started | 38 (All patients that received treatment went into follow up period.)
Completed | 26
Not Completed | 12
Not completed — Other | 12

BASELINE CHARACTERISTICS:
Population: Patients that completed induction of capecitabine and oxaliplatin, were then enrolled and completed treatment in capecitabine, oxaliplatin, and radiation.
Arm/Group | Induction and Combination Treatment
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Determine Pathologic Complete Response
Description: Pathologic response will be assessed semiquantitatively irrespective of lymph node status based on the estimated percentage of residual carcinoma in relation total carcinoma area, including amount of radiotherapy-induced tissue injury, in mural histologic sections.
  Pathologic response will be defined as:
  P0: 0% residual cancer P1: 1% to 50% residual cancer P2: more than 50% residual cancer
Time Frame: At time of surgery
Population: Patients analyzed were patients that reached and completed surgery.
Measure: Count of Participants; unit: Participants
Groups:
- Induction, Combination and Surgery: Induction Therapy: Two 21-day cycles will be given as induction. Weeks 1-6:
  Capecitabine will be given at 1000 mg/m2 twice daily approximately 12 hours apart for 14 days, followed by seven days off.
  Oxaliplatin will be given at 70 mg/m2 intravenously in 5% dextrose over 2 hours on days 1 and 8 of each cycle.
  Combination Therapy: Two 21-day cycles will be given for combination therapy Weeks 7-12:
  Capecitabine will be given at 825 mg/m2 twice daily approximately 12 hours apart for five days (Monday through Friday) followed by two days off for 51/2 weeks.
  Oxaliplatin will be given at 50 mg/m2 intravenously in 5% dextrose over two hours on days 1, 8 and 15 of each cycle.
  Radiation: 1.8 Gy daily Monday through Friday to a total of 50.4 Gy for 6 weeks during combination therapy.
  4-6 weeks later subjects will undergo evaluation for response and surgical resection.
Arm/Group | Induction, Combination and Surgery
Number analyzed (Participants) | 28
Participants | 9

2. Secondary Outcome: Clinical Response Rate
Description: Clinical response Rate will be expressed as the proportion of patients demonstrating a complete and/or partial response based on all evaluable patients treated.Clinical response will be evaluated according to Response Evaluation Criteria In Solid Tumors 1.0 (RECIST) .
  Complete Response (CR) is defined as the disappearance of all target lesions Partial Response (PR) is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions,taking as reference the baseline sum LD
Time Frame: four to six weeks following completion of 4 cycles (1 cycle = 21days) of chemotherapy treatment and prior to surgery
Population: 1 patient was registered to the study but was not treated on study and was therefore not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction and Combination Treatment
Number analyzed (Participants) | 43
Participants | 28

3. Secondary Outcome: Recurrence Rate
Description: Recurrence rate will be defined as disease recurrence, progressive disease or death. Patients will be followed for disease recurrence or death until the end of the study.
Time Frame: From the time of start of treatment until first documentation of disease recurrence, progression or death, whichever comes first until the end of the study, a maximum of 6 years and 7 months.
Population: 1 patient was registered but not treated on study and therefore was not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction and Combination Treatment
Number analyzed (Participants) | 43
Participants | 23

4. Secondary Outcome: Time to Progression
Description: Time to Progression will be measured as time from the first day of therapy until death, disease progression or last contact.
Time Frame: From start of first treatment until time of first documentation of progression of disease or death, whichever comes first, until the study closes, up to a maximum of 6 years and 7 months.
Population: Data collected was not analyzed before the study was terminated. Count of participants indicates the number of patients with progressive disease or death at the time the study closed permanently.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction, Combination and Surgery
Number analyzed (Participants) | 43
Participants | 28

5. Secondary Outcome: Patterns of Failure
Time Frame: At time of surgery
Population: No data collected for this outcome measure. There is no data to report on.
Arm/Group | Induction and Combination Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Toxicity Profile
Description: Toxicity will be assessed at the beginning of every cycle during chemotherapy for a total of 4 cycles (1 cycle =21 days) and then 30 days post last dose of chemotherapy. All toxicities will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 (CTCAE 3.0)
  In general adverse events (AEs) will be graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
  Only incidents of AEs determined to be related to chemotherapy are recorded here.
Time Frame: During chemotherapy treatment and up to 30 days post-last dose of chemotherapy.
Population: Toxicity data was collected and analysed for the first 40 patients.
Measure: Number; unit: participants
Arm/Group | Induction and Combination Treatment
Number analyzed (Participants) | 40
participants
  Thrombocytopenia | 20
  Anemia | 17
  lymphopenia | 16
  Leukopenia | 15
  Neutropenia | 8
  Thrombosis | 5
  Nausea | 18
  Diarrhea | 15
  Dysphagia | 15
  Vomiting | 8
  Constipatation | 7
  Abdominal pain | 6
  Stomatitis | 6
  Esophgitis | 4

7. Secondary Outcome: Correlate Proteomic and Pharmacologic Characteristics With Prognosis and Response to Therapy.
Time Frame: At time of sugery
Population: No data was collected for this outcome measure. There is no data to report on.
Arm/Group | Induction and Combination Treatment
Number analyzed (Participants) | 0

8. Post Hoc Outcome: Determine Progressive Free Survival
Time Frame: After cycles 2, and 4 (pre-surgery) 30 days after surgery and then every 3 months until first documentation of progressive disease, death and up to a maximum of 24 months.
Population: The only data collected for this outcome measure was progression free survival rate at 3 months, 6 months, and 12 months.
Measure: Number; unit: percentage of patents progression free
Arm/Group | Induction and Combination Treatment
Number analyzed (Participants) | 43
percentage of patents progression free
  3 months | 86.05
  6 months | 67.44
  12 months | 62.62
  24 months | 51.83

9. Post Hoc Outcome: Overall Survival
Time Frame: From the start of treatment and then every 3 months until death or a maximum of 24 months.
Population: 1 patient was registered to the study, but was not treated on study and was therefore not evaluable. Data for overall surivival was collected at 3 months, 6 months, 12 months and 24 months. There was no further data analysis completed
Measure: Number; unit: percentage of patients alive
Arm/Group | Induction and Combination Treatment
Number analyzed (Participants) | 43
percentage of patients alive
  3 months | 93.02
  6 months | 83.72
  12 months | 66.81
  24 months | 58.51

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 6 years, 7 months.
Description: For this study, only adverse events of the highest grade that were considered clinically significant were collected. Only serious adverse event that are fatal or life-threatening (i.e., results in an immediate risk of death), is permanently or substantially disabling, requires or prolongs hospitalization (only of related to an unexpected complication), or is a congenital anomaly, new cancer or medication overdose, or that the investigator deemed important were collected.
Arm/Group | Induction and Combination Treatment
All-Cause Mortality (participants affected / at risk) | 28/44
Serious Adverse Events (participants affected / at risk) | 10/43
Other Adverse Events (participants affected / at risk) | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction and Combination Treatment (N=43)
Supraventricular and nodal arrhythmia:Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Cardiac general:Congestive heart failure (Cardiac disorders) | 1 (1)
CARDIAC ARRHYTHMIA: Cardiac arrest (Supraventricular and nodal arrhythmia: Atrial fibrillation) (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1)
Cellulitis (skin infection) (Infections and infestations) | 1 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Suicide (Social circumstances) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction and Combination Treatment (N=43)
Hemoglobin (Anemia) (Blood and lymphatic system disorders) | 24 (24)
Neutrophils (Neutropenia) (Blood and lymphatic system disorders) | 8 (8)
Leukocytes (total white blood count) (Blood and lymphatic system disorders) | 22 (22)
Lymphopenia (Blood and lymphatic system disorders) | 20 (20)
Platelets (Thrombocytopenia) (Blood and lymphatic system disorders) | 28 (28)
Hypotension (Cardiac disorders) | 8 (8)
Palpitations (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia: multifocal atrial tachycardia (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia:Tachycardia (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 33 (33)
Fever (General disorders) | 6 (6)
Insomnia (General disorders) | 3 (3)
Rigors (General disorders) | 1 (1)
Sweating (General disorders) | 2 (2)
Weight loss (General disorders) | 14 (14)
cardiac (Cardiac disorders) | 1 (1)
(International Normalized Ratio of prothrombin time) (Investigations) | 2 (2)
Skin (Skin and subcutaneous tissue disorders) | 12 (12)
Anorexia (Gastrointestinal disorders) | 17 (17)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 11 (11)
Colitis (Gastrointestinal disorders) | 4 (4)
Dehydration (Gastrointestinal disorders) | 15 (15)
Diarrhea (Gastrointestinal disorders) | 22 (22)
Esophagitis (Gastrointestinal disorders) | 6 (6)
Mucositis/Stomatitis (Gastrointestinal disorders) | 10 (10)
Heartburn (dyspepsia) (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 28 (28)
Vomiting (Gastrointestinal disorders) | 17 (17)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Difficulty swallowing (dysphagia) (Gastrointestinal disorders) | 16 (16)
Nose bleed (General disorders) | 3 (3)
Infection (not otherwise specified) (Infections and infestations) | 4 (4)
Colitis, infectious (Infections and infestations) | 1 (1)
Pulmonary infection (Infections and infestations) | 1 (1)
Upper airway infection (not otherwise specified) (Infections and infestations) | 1 (1)
Infection (Sepsis) (Infections and infestations) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Alkaline phosphatase (increase) (Metabolism and nutrition disorders) | 5 (5)
ALT/SGPT - serum glutamic pyruvic transaminase (increase) (Metabolism and nutrition disorders) | 5 (5)
AST/SGOT -serum glutamic oxaloacetic transaminase (increase) (Metabolism and nutrition disorders) | 7 (7)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4 (4)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 5 (5)
Creatinine (increase) (Metabolism and nutrition disorders) | 3 (3)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 10 (10)
Potassium, serum-low(hypokalemia) (Metabolism and nutrition disorders) | 6 (6)
Sodium, serum-low(hyponatremia) (Metabolism and nutrition disorders) | 3 (3)
Neuropathy: motor (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 27 (27)
Confusion (Psychiatric disorders) | 2 (2)
Dizziness (Psychiatric disorders) | 2 (2)
Cold sensitivity (Nervous system disorders) | 1 (1)
Mood alteration - Depression (Psychiatric disorders) | 2 (2)
Esophagus pain (Gastrointestinal disorders) | 4 (4)
Abdomen pain (Not otherwise specified) (Gastrointestinal disorders) | 7 (7)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Jaw pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain NOS (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain swallowing (Odynophagia) (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Shortness of breath (dyspnea) (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes